CLINICAL TRIAL: NCT03103477
Title: Platelet Activating Factor Stability in Urine
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Eugen C. Campian, MD, Principal investigator, St. Louis University
Other Study IDs: 27756
Record Dates: First submitted 2017-01-18; First posted 2017-04-06 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study is proposing to assess PAF and PAF-AH activity in urine after using various handling methods of the urine specimen. Better understanding of PAF stability will allow for better design of future experiments involving PAF in interstitial cystitis patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Office: Patients presenting for a routine office visit will be asked to donate at least 50 ml of urine. The urine specimen will be aliquoted in containers, one with and one without a PAF-AH inhibitor and kept at room temperature.
  The aliquots (2mL) will be frozen at predetermined intervals of 5, 10, 20, 40 and 60 min from time of collection in liquid nitrogen and then later stored in -80 freezer.
  Interventions: Other: Urine stability
- Surgery: A separate group of patients undergoing surgery lasting more than 60 min operating time, will be consented as well. These patients have Foley catheters in place during the surgery. Five cc's of urine will be collected from the catheter at pre-determined intervals 5, 10, 20, 40 and 60 minutes, aliquoted (2mL) and frozen in liquid nitrogen and later stored in the -80 freezer.
  Interventions: Other: Urine stability

INTERVENTIONS:
Other: Urine stability — This study is proposing to assess PAF and PAF-AH activity in urine after using various handling methods of the urine specimen. Better understanding of PAF stability will allow for better design of future experiments involving PAF in interstitial cystitis patients.

SUMMARY:
The investigator's hypothesis is that smoking induces inflammation in the bladder wall. This may predispose to the development of Interstitial cystitis(IC) / bladder pain syndrome(BPS). Previous research has linked one the Platelet Activating Factor - PAF to interstitial cystitis. The investigators will study a limited number of patients to determine whether PAF is stable in urine and whether special precautions (for example - immediate freezing in liquid nitrogen) is necessary for accurate measurement of PAF in the urine.

Patients who are presenting for an office visit will be asked to donate at least 50 ml of urine.

A separate group of patients who are scheduled for surgery, are also being asked to donate around 25 ml of urine during surgery.

No patient data other than group assignment, whether they smoke or if they have or not have interstitial cystitis will be recorded.

DETAILED DESCRIPTION:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a severe, chronic bladder condition that is extremely painful and disruptive. Incidence of the disease has increased dramatically in recent years, primarily due to enhanced awareness and better defined inclusion criteria. Difficulty in diagnosis arises from the diversity of symptoms and severity between patients and in the same patient at different times. IC/BPS is generally accepted as a disease of exclusion in which a diagnosis is reached after ruling out other conditions. A firm diagnosis is only mildly assuring for patients because there are very few therapeutic approaches that can alleviate the symptoms. Several risk factors are associated with IC/BPS, including age, sex and race [5] and modifiable risk factors such as diet and smoking. This proposal is to test the hypothesis that cigarette smoking contributes directly to changes in the bladder that are indicative of, or predispose to, IC/BPS. In preliminary studies, the investigators have exposed mice to cigarette smoke and observed breaks in the urothelium, decreased urothelial tight junction protein expression, increased vascularity and inflammatory cells in the bladder wall. This lab has previously demonstrated that cigarette smoke inhibits endothelial cell platelet activating factor acetylhydrolase (PAF-AH), which is responsible for the hydrolysis of PAF, resulting in increased PAF, a membrane phospholipid-derived inflammatory mediator. The investigators have also shown that calcium-independent phospholipase A2β (iPLA2β) is responsible for the majority of PAF production in endothelial and urothelial cells. PAF has been shown to increase matrix metalloproteinases (MMP) which in turn inhibit anti-angiogenic pigment epithelium-derived factor (PEDF), thus promoting angiogenesis. These studies indicate a direct relationship between PAF accumulation and PEDF expression in the bladder that may contribute to inflammation in smokers.

PAF stability in urine has not been established in the literature. This study is proposing to assess PAF and PAF-AH activity in urine after using various handling methods of the urine specimen. Better understanding of PAF stability will allow for better design of future experiments involving PAF in interstitial cystitis patients.

The investigators have exposed mice to cigarette smoke and examined changes in the bladder. they have observed thinning and sloughing of the urothelium, plus increased vascularization. These changes are observed in the bladder wall of IC/BPS patients. We have measured increased PAF accumulation and decreased expression of PEDF in the bladder wall.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting for routine care in the UroGynecology division or
* Patient undergoing gynecologic or urogynecologic surgery exceeding 60 minute operating time.

Exclusion Criteria:

* Age less than 18 or more than 80
* Unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult females with r without IC
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
PAF production | 1 hour
  elicits changes in the bladder wall that can predispose to IC/BPS. In this aim, the investigators will determine whether urine PAF is stable at room temperature, or whether special precautions (e.g. freezing or use of PAF-AH inhibitors) are needed for accurate PAF measurements in urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Eugen C Campian, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No